CLINICAL TRIAL: NCT06897904
Title: Basic Hematological Parameters and Coagulation Profile in Type 1 Diabetic Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramez Nady Kamel Ragheb, Residant doctor, Assiut University
Other Study IDs: hemo& coag type 1 DM
Record Dates: First submitted 2025-03-15; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- diabetic group: type 1 diabetic children
- control group: healthy control

SUMMARY:
Diabetes mellitus is a group of chronic metabolic diseases characterized by hyperglycemia .Type 1 diabetes is a heterogeneous disease related to the destruction of pancreatic beta cells and is a result of absolute lack of insulin

* Diabetes mellitus has been traditionally looked upon as a disease of adults (except Type I diabetes), however it can affect individuals of any age. Given the peculiarities and problems that it carries, diabetes in children and adolescents poses special challenges to the entire society. Diabetes is the second commonest chronic disease occurring in 1 in every 1500 children by age 5 and in 1 in 350 children by age 8 . Microvascular (retinopathy, neuropathy, and nephropathy) Aim of the research to assess basic hematological parameters and coagulation profiles among type 1 diabetic children and compare them with healthy controls and macrovascular (coronary artery disease, peripheral vascular disease, and cerebrovascular disease) atherothrombotic complications may occur in children and adolescents, depending on the duration of diabetes, the degree of metabolic control, and other factorssuch as genetics . Diabetes mellitus can cause blood disorders such as deformity of red blood cells and increase their adhesion [6].It has an effect on the function of red blood cells through the interaction with the membrane and intracellular components . Red blood cell distribution width (RDW) is a measure of the difference in the size of red blood cells. An increase in RDW can be caused by anemia or nutritional deficiencies related to anemia
* Studies have shown that the average number of red blood cells, hemoglobin and hematocrit in diabetic patients is lower than the control group, which indicates the presence of anemia in diabetic patients .

ELIGIBILITY:
Inclusion Criteria:

* Age from one month to 18 year.
* Both sexes.
* Patients known to have type 1 diabetes.

Exclusion Criteria:

* Patients less than one month and more than 18years.
* history of bleeding disorders or anemia unrelated to diabetes.
* Otherc types of diabetes .

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: type 1 diabetic children and matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Prothrombin time | baseline
  comparison of prothrombin time between T1DM children and healthy controls